CLINICAL TRIAL: NCT04693715
Title: RESCUE: A Randomized, Blinded, Placebo-controlled, Parallel Group Design to Determine the Safety of RNS60 in Large Vessel Occlusion Stroke Patients Undergoing Endovascular Thrombectomy
Brief Title: Safety of RNS60 in Large Vessel Occlusion Stroke Patients Undergoing Endovascular Thrombectomy
Acronym: RESCUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06.5.1.H1
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Ischemic
Keywords: Endovascular Thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — RNS60

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RNS60 0.5 mL/kg/h (Experimental): RNS60 0.5 mL/kg/h infusion for 48h (up to a maximum of 65 mL/h) starting within 30 min of randomization (but prior to arterial access closure)
  Interventions: Drug: RNS60
- RNS60 1.0 mL/kg/h (Experimental): RNS60 1.0 mL/kg/h infusion for 48h (up to a maximum of 130 mL/h) starting within 30 min of randomization (but prior to arterial access closure)
  Interventions: Drug: RNS60
- Placebo 1.0 mL/kg/h (Placebo Comparator): Placebo (normal saline) 1.0 mL/kg/h infusion for 48h (up to a maximum of 130 mL/h) starting within 30 min of randomization (but prior to arterial access closure)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RNS60 — RNS60 injection solution
  Arms: RNS60 0.5 mL/kg/h; RNS60 1.0 mL/kg/h
Drug: Placebo — Placebo injection solution
  Arms: Placebo 1.0 mL/kg/h

SUMMARY:
A Phase II, randomized, blinded, placebo-controlled, parallel group study with patients experiencing a large vessel occlusion acute ischemic stroke who are selected for endovascular revascularization. Participants will be given a 48 h infusion of either 0.5 mL/kg/h RNS60 (up to a maximum of 65 mL/h), 1.0 mL/kg/h RNS60 (up to a maximum of 130 mL/h), or 1.0 mL/kg/h (up to a maximum of 130 mL/h) placebo (normal saline) starting within 30 minutes of consent after confirmation of candidacy for endovascular thrombectomy.

DETAILED DESCRIPTION:
This study is a Phase II, randomized, blinded, placebo-controlled, parallel group design. Participants experiencing a large vessel occlusion acute ischemic stroke who are selected for endovascular revascularization will be given a 48 h infusion of either 0.5 mL/kg/h RNS60 (up to a maximum of 65 mL/h), 1.0 mL/kg/h RNS60 (up to a maximum of 130 mL/h), or 1.0 mL/kg/h (up to a maximum of 130 mL/h) placebo (normal saline) starting within 30 minutes of consent after confirmation of candidacy for endovascular thrombectomy and prior to arterial closure. Outcomes of the main trial will be evaluated throughout a 90 day observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke (AIS) selected for emergency endovascular treatment.
2. Age 18 years or older.
3. Onset (last-known-well) time to randomization time within 24 hours.
4. Disabling stroke defined as a baseline National Institutes of Health Stroke Score (NIHSS)

   1. NIHSS > 5 for internal carotid artery (ICA) and M1-middle cerebral artery (MCA) occlusion or
   2. NIHSS > 10 for M2-MCA occlusion.
5. Confirmed symptomatic intracranial occlusion at one or more of the following locations: Intracranial carotid I/T/L, M1 or M2 segment MCA. Tandem extracranial carotid and intracranial occlusions are permitted.
6. Pre-stroke (24 hours prior to stroke onset) historical modified Rankin Scale (mRS) ≤2. Patient must be living independently without requiring nursing care.
7. Qualifying imaging performed less than 2 hours prior to randomization.
8. Consent process completed as per applicable laws and regulation and the IRB requirements.

Exclusion Criteria:

1. Evidence of a large core of established infarction defined as Alberta Stroke Program Early Computerized Tomography Score (ASPECTS) 0-4.
2. Evidence of absence of collateral circulation on qualifying imaging (collateral score of 0 or 1 if multiphase computed tomography angiography (mCTA) is used, or absence of adequate ischemic penumbra in the judgment of the Investigator if computed tomographic perfusion (CTP) is used).
3. Any evidence of intracranial hemorrhage or mass lesion on the qualifying imaging.
4. Planned use of an endovascular device not having approval or clearance by the relevant regulatory authority.
5. Endovascular thrombectomy procedure is completed as defined by the presence of arterial access closure.
6. Clinical history, past imaging or clinical judgment suggesting that the intracranial occlusion is chronic or there is suspected intracranial dissection such that there is a predicted lack of success with endovascular intervention.
7. Estimated or known weight > 130 kg (287 lbs).
8. Known pregnant/lactating female.
9. Myocardial infarction (MI) within 6 months prior to Screening including non-Q wave MI; Diagnosis of congestive heart failure (CHF) with either:

   1. current clinical signs and symptoms of ventricular dysfunction (e.g., edema, shortness of breath),
   2. CHF medication adjustment within the prior 30 days or
   3. ejection fraction (if report available) of 30% or less measured in the 6 months prior to Screening; as either medically documented or reported by patient or another person considered by the Investigator to be reasonably reliable.
10. Known renal impairment defined as requiring renal replacement therapy (hemo- or peritoneal dialysis).
11. Inability to have magnetic resonance imaging (MRI) (Non-magnetic resonance [MR] compatible implants or any other foreseeable reason, including claustrophobia)
12. Severe or fatal comorbid illness that will prevent improvement or follow up.
13. Inability to complete follow-up treatment to Day 90.
14. Participation in another clinical trial investigating a drug, medical device, or a medical procedure in the 30 days preceding trial inclusion and throughout the duration of the trial.
15. Reported known seizure at time of stroke onset.
16. Ischemic stroke within previous 30 days.
17. Patients in normal sinus rhythm with a known QTcF > 460 ms at Screening.
18. Any other symptom that in the investigator's opinion may complicate or preclude the subject from participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Northwestern University, Chicago, Illinois
  - Oregon Health & Science University, Portland, Oregon
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghosh S, Dubow JS, Sutherland J, Smith W, Chiu D, Clark WM, Favilla CG, Ansari SA, Kalmes A, Mock J, Cook DJ, Madsen TE, Jayaraman M, Moldovan K, Torabi R, Liebeskind DS, Fisher M, McTaggart RA. Randomized, Proof-of-Concept Trial (RESCUE) of RNS60 as an Adjunct Therapy in Acute Ischemic Stroke. Stroke. 2025 Sep;56(9):2386-2397. doi: 10.1161/STROKEAHA.125.051179. Epub 2025 Jul 17. PMID 40671649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 sites in the United States.
Pre-assignment Details: Participants experiencing a large vessel occlusion (LVO) acute ischemic stroke (AIS) who were selected for endovascular thrombectomy (EVT) were randomized in a 1:1:1 ratio to one of three arms in the study. Participants were given a 48-hour infusion of either 0.5 milliliter/kilogram/hour (mL/kg/h) RNS60, 1.0 mL/kg/h RNS60, or 1.0 mL/kg/h placebo (normal saline).
Groups:
- RNS60 1.0 mL/kg/h: Participants received RNS60 1.0 mL/kg/h infusion for 48 hours (up to a maximum of 130 mL/h) starting within 30 min of randomization (but prior to arterial access closure).
- RNS60 0.5 mL/kg/h: Participants received RNS60 0.5 mL/kg/h infusion for 48 hours (up to a maximum of 65 mL/h) starting within 30 min of randomization (but prior to arterial access closure).
- Placebo 1.0 mL/kg/h: Participants received placebo (normal saline) 1.0 mL/kg/h infusion for 48 hours (up to a maximum of 130 mL/h) starting within 30 min of randomization (but prior to arterial access closure).
Period: Overall Study
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Started | 24 | 31 | 28
Intent-to-treat (ITT) Population (ITT Population: All randomized participants who received study drug regardless of treatment actually received.) | 24 | 30 | 28
Safety Population (Safety Population: All randomized participants who received any volume of study drug based on the actual treatment received.) | 24 | 30 | 28
Completed | 22 | 25 | 21
Not Completed | 2 | 6 | 7
Not completed — Adverse Events Leading to Death | 2 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Legal Authorized Representative | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population: All randomized participants who received study drug regardless of treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h | Total
Number analyzed (Participants) | 24 | 30 | 28 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (10.65) | 68.0 (12.51) | 66.0 (12.50) | 67.2 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 11 | 31
  Male | 17 | 17 | 17 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 22 | 28 | 27 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 21 | 23 | 24 | 68
    Black or African American | 2 | 6 | 1 | 9
    Asian | 1 | 1 | 2 | 4
    Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or resulted in a congenital anomaly/birth defect. An SAE could also be an important medical event that may not have resulted in death, was life-threatening, or required hospitalization, but jeopardized the participant and required medical or surgical intervention to prevent one of the outcomes listed above. Treatment-emergent SAEs were defined as SAEs that started after the start of study drug infusion and are reported here.
Time Frame: From start of study drug administration up to Day 90
Population: Safety Population: All randomized participants who received any volume of study drug based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 24 | 30 | 28
Participants | 6 | 10 | 8

2. Primary Outcome: Mortality: Proportion of Participants Alive at Day 90
Time Frame: Day 90
Population: ITT Population: All randomized participants who received study drug regardless of treatment actually received.
Measure: Number; unit: proportion of participants
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 24 | 30 | 28
proportion of participants | 0.917 | 0.933 | 0.857

3. Secondary Outcome: Number of Participants With Non-disability Based on Modified Rankin Scale (mRS ) Score at Day 90
Description: The mRS is a clinician-reported outcome measure for participants who have suffered a stroke. It measures functional recovery as the degree of disability or dependence in daily activities in a 6-point disability scale with possible scores ranging from 0 to 5: 0-no symptoms at all; 1-no significant disability despite symptoms; able to carry out all usual duties and activities; 2-slight disability: unable to carry out all previous activities but able to look after own affairs without assistance; 3-moderate disability: requiring some help, but able to walk without assistance; 4-moderately severe disability: unable to walk without assistance and unable to attend to own bodily needs without assistance; 5-severe disability; bedridden, incontinent, requiring constant nursing care and attention. A score of 6 is used for participants who expire (death). Non-disability was defined as a score ranging from 0 to 2. Disability was defined as a score ranging from 3-6.
Time Frame: Day 90
Population: ITT Population: All randomized participants who received study drug regardless of treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 24 | 30 | 28
Participants | 15 | 13 | 13

4. Secondary Outcome: Change From Baseline in Infarct Volume of Stroke at 48 Hours
Description: Infarct progression/regression was measured by Magnetic Resonance Imaging (MRI) of the brain. The mean change from post-EVT baseline in the volume of injured tissue was calculated at 48 hours.
Time Frame: Baseline, 48 hours
Population: ITT Population: All randomized participants who received study drug regardless of treatment actually received. Number of participants analyzed is the number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 24 | 29 | 28
mL
  Baseline | 43.6 (40.26) [0.9 to 137.8] | 37.9 (41.82) [0.0 to 175.6] | 49.0 (55.93) [1.2 to 213.9]
  Change From Baseline at 48 Hours: number analyzed (Participants) | 23 | 26 | 27
  Change From Baseline at 48 Hours | 21.4 (23.16) [0.2 to 86.6] | 27.1 (30.00) [-1.6 to 84.8] | 40.6 (42.20) [1.1 to 172.6]

5. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS) at 24 Hours
Description: The NIHSS is a standardized neurological examination scale that is a measure of disability and recovery after acute stroke. The NIHSS assessment is a standardized 15-item impairment scale intended to evaluate neurologic outcome and degrees of recovery for subjects with stroke. The scale assesses levels of consciousness, extraocular movements, visual fields, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect). The NIHSS was scored by those trained in the use of this scale. Each item was scored in ranges 0-2, 0-3, or 0-4. A score of 0 indicates normal performance. Total scores on the NIHSS ranged from 0-42, with higher values reflecting increasing severity. Stroke severity was further stratified in the following way: > 25: Very severe; 15-24: Severe; 5-14: Mild to moderately severe; < 5: Mild.
Time Frame: 24 hours
Population: ITT Population: All randomized participants who received study drug regardless of treatment actually received. The number of participants analyzed is the number of participants with data available at the 24 hour time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 24 | 29 | 27
score on a scale | 8.3 (6.77) | 10.4 (7.67) | 10.9 (7.88)

6. Secondary Outcome: Proportion of Participants With Worsening of Stroke
Description: Worsening of stroke was defined as progression, or hemorrhagic transformation of the index stroke, as documented by brain imaging, which is (a) life-threatening requiring intervention and/or (b) results in increased disability as gauged by a ≥ 4-point increase from lowest NIHSS pre-decline and/or (c) results in death. Proportion of participants with worsening of stroke was calculated as number of participants with worsening of stroke divided by the total number of participants observed over the 90-day period in each arm.
Time Frame: Up to Day 90
Population: ITT Population: All randomized participants who received study drug regardless of treatment actually received.
Measure: Number; unit: proportion of participants
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 24 | 30 | 28
proportion of participants | 0.208 | 0.400 | 0.286

7. Secondary Outcome: Percentage of Participants With Barthel Index (BI) Score ≥95 at Day 90
Description: The BI is an index of functional independence. Its values range from 0 to 100, with higher scores indicating greater independence. Score range in BI items: Feeding 0-10; Bathing 0-5; Grooming 0-5; Dressing 0-10; Bowels 0-10; Bladder 0-10; Toilet use 0-10; Transfers (bed to chair and back) 0-15; Mobility (on level surfaces) 0-15; Stairs 0-10. Item scores vary in increments of 5 points. Functional independence at Day 90 was evaluated. Participants having a score ≥95 on the BI Score were deemed to have achieved functional independence, whereas those scoring <95 at Day 90 were deemed to have failed to achieve functional independence.
Time Frame: Day 90
Measure: Number; unit: percentage of participants
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 24 | 30 | 28
percentage of participants | 70.8 | 40.0 | 42.9

8. Secondary Outcome: Health-related Quality of Life as Measured by 5-Level EuroQoL 5D Index (EQ-5D-5L) at Day 90
Description: EQ-5D-5L is a generic instrument for measuring health-related quality of life. It consists of a 5-item questionnaire, which was interviewer administered by study staff. The 5-item questionnaire comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and each dimension has 5 response levels (1-no problems, 2-slight problems, 3-moderate problems, 4-severe problems, 5-unable to/extreme problems). The health state is then summarized to be a single number, EQ-5D-5L Index score, by applying a country-specific standard value set. EQ-5D-5L Index score for the United States ranges from -0.59 to 1, where 1 indicates a better health condition.
Time Frame: Day 90
Population: ITT Population: All randomized participants who received study drug regardless of treatment actually received. Number of participants analyzed is the number of participants with available data on Day 90.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
Number analyzed (Participants) | 21 | 23 | 19
score on a scale | 0.77 (0.29) | 0.60 (0.33) | 0.66 (0.28)

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to Day 90
Description: Treatment-emergent AEs were defined as AEs that started after the start of study drug infusion and are reported here. Safety Population: All randomized participants who received any volume of study drug based on the actual treatment received.
Arm/Group | RNS60 1.0 mL/kg/h | RNS60 0.5 mL/kg/h | Placebo 1.0 mL/kg/h
All-Cause Mortality (participants affected / at risk) | 2/24 | 2/30 | 4/28
Serious Adverse Events (participants affected / at risk) | 6/24 | 10/30 | 8/28
Other Adverse Events (participants affected / at risk) | 21/24 | 28/30 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RNS60 1.0 mL/kg/h (N=24) | RNS60 0.5 mL/kg/h (N=30) | Placebo 1.0 mL/kg/h (N=28)
Stroke in evolution (Nervous system disorders) | 1 | 2 | 3
Brain edema (Nervous system disorders) | 0 | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 0 | 1 | 0
Hemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Bacteremia (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Klebsiella bacteremia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral ischemia (Vascular disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RNS60 1.0 mL/kg/h (N=24) | RNS60 0.5 mL/kg/h (N=30) | Placebo 1.0 mL/kg/h (N=28)
Headache (Nervous system disorders) | 9 | 3 | 4
Hemorrhagic transformation stroke (Nervous system disorders) | 2 | 1 | 5
Stroke in evolution (Nervous system disorders) | 2 | 2 | 2
Subarachnoid hemorrhage (Nervous system disorders) | 2 | 1 | 3
Brain edema (Nervous system disorders) | 2 | 0 | 3
Cerebral hemorrhage (Nervous system disorders) | 1 | 2 | 2
Neuralgia (Nervous system disorders) | 0 | 3 | 0
Brain compression (Nervous system disorders) | 2 | 0 | 0
Cerebral mass effect (Nervous system disorders) | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 2 | 0
Hemorrhagic cerebral infarction (Nervous system disorders) | 2 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 8 | 6 | 7
Dysphagia (Gastrointestinal disorders) | 3 | 5 | 3
Anal incontinence (Gastrointestinal disorders) | 2 | 3 | 4
Nausea (Gastrointestinal disorders) | 3 | 4 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 0 | 3
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 5 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 4 | 4
Acute kidney injury (Renal and urinary disorders) | 1 | 3 | 2
Incontinence (Renal and urinary disorders) | 0 | 1 | 3
Hematuria (Renal and urinary disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 5 | 3 | 4
Hypertension (Vascular disorders) | 0 | 2 | 3
Deep vein thrombosis (Vascular disorders) | 2 | 2 | 0
Peripheral artery occlusion (Vascular disorders) | 2 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 6 | 2
COVID-19 (Infections and infestations) | 1 | 3 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 4 | 4
Bradycardia (Cardiac disorders) | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 3 | 4 | 3
Agitation (Psychiatric disorders) | 2 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 1 | 2
Ejection fraction decreased (Investigations) | 0 | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2
Dry eye (Eye disorders) | 0 | 2 | 2
Pyrexia (General disorders) | 0 | 3 | 1
Gastrostomy (Surgical and medical procedures) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only a) after first publication of the data by the sponsor or b) 18 months after the study has been completed, whichever comes first. The sponsor can review results communications 30 days prior to public release and can delay these for no more than 60 days from the date that the request is given to the investigator. The sponsor cannot require changes to the communication, other than to remove sponsor confidential information, and cannot unilaterally extend the delay.

DOCUMENTS (2):
  • Study Protocol (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT04693715/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04693715/SAP_001.pdf